CLINICAL TRIAL: NCT07163975
Title: Success of Complete Pulpotomy and Root Canal Treatment and Quality of Life in Patients With Symptomatic Irreversible Pulpitis With Type 2 Diabetes Mellitus: A Randomized Clinical Trial
Brief Title: Complete Pulpotomy and Root Canal Treatment Patients With Irreversible Pulpitis With Type 2 Diabetes Mellitus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Anmol Jain
Record Dates: First submitted 2025-08-25; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-04

CONDITIONS: Type 2 Diabetes Mellitus (T2DM); Irreversible Pulpitis
Keywords: pulpotomy; type 2 Diabetes Mellitus; irreversible pulpitis
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- complete pulpotomy (Experimental): complete pulpotomy will be performed in teeth with irreversible pulpitis in diabetic patients.
  Interventions: Procedure: complete pulpotomy
- Root Canal Treatment (Active Comparator): root canal treatment will be performed in teeth with irreversible pulpitis in diabetic patients.
  Interventions: Procedure: Root canal treatment

INTERVENTIONS:
Procedure: complete pulpotomy — the exposed pulp tissue will be amputated using fresh sterile large round diamond bur in a high-speed hand-piece under water coolant to the level of canal orifices. The pulp wound will be irrigated with 3% NaOCl. For hemostasis, sterile cotton soaked in 3% NaOCl will be placed over the pulpal wound for 2 minutes, repeated for up to 5 min if required. Root canal therapy will be initiated in cases in which haemostasis is not achieved within 5 minutes. After hemostasis, MTA will be placed in thickness of 2 to 3 mm over the pulp exposure site using a carrier. This will be followed by application of a layer of light-cure RMGIC and light-curing for 20 sec. The tooth then will be restored using composite resin following etch and rinse technique.
  Arms: complete pulpotomy
Procedure: Root canal treatment — RCT will be performed in single visit. Root canal orifices will be explored using a DG 16 probe. A size 10 or 15 K-file will be passively inserted into the coronal two- thirds of the canal to verify a smooth glide path.
  Coronal enlargement will be done using Gates-Glidden drills. Working length will be determined with the help of electronic apex locator and will be confirmed radiographically. Canals will be prepared using the crown down technique with NiTi rotary instruments. The master apical file (MAF) size for each canal will be selected to be three sizes larger than the initial apical binding file at the WL. 5ml of 5.25% sodium hypochlorite using a 30-gauge side-vented needle will be used for optimal irrigation after each instrument.
  After completion of canal instrumentation, the canals will be irrigated with 5.0 ml of 17% ethylene-diamine-tetra acetic acid for 1 minute followed by a final irrigation with 5.0 ml of 5.25% sodium hypochlorite. Canals will be dried with
  Arms: Root Canal Treatment

SUMMARY:
there is limited endodontic research on the effects of DM on pulp tissues. Diabetic human and animal histological research have demonstrated decreased wound repair, chronic pulp inflammation and reduced dentin bridge formation. To date, no human clinical trial has examined the impact of diabetes mellitus on teeth with irreversible pulpitis. Due to the paucity of data in the literature, there is a clinical dilemma whether to recommend root canal therapy or vital pulp therapy in diabetic patients with irreversible pulpitis.

To the best of our knowledge, no prospective study has evaluated the outcome of complete pulpotomy versus root canal treatment in T2DM patients with irreversible pulpitis. The aim of this study is to compare and evaluate the success rates of pulpotomy and root canal treatment in type 2 diabetes mellitus patients in mature permanent teeth presenting with clinical symptoms of irreversible pulpitis.

DETAILED DESCRIPTION:
Rationale: - Preservation of pulp vitality is a critical factor in long-term tooth survival. In extremely deep carious lesion with symptomatic irreversible pulpitis, vital pulp therapy procedures in the form of complete pulpotomy is a more conservative treatment strategy, based on the premise that a biologically active material placed in direct contact with the pulp wound can determine the pulpal response and result in the development of a reparative hard tissue bridge to preserve pulp vitality. Scientific literature indicates that type 2 diabetes mellitus has a detrimental effect on the wound healing capacity of dental pulp, however lacks evidence in clinical studies. to the best of our knowledge no study has been done till date comparing the outcome of complete pulpotomy and root canal treatment in patients with type 2 diabetes mellitus with clinical signs of irreversible pulpitis.

Aim- To compare the outcome of complete pulpotomy and root canal treatment in mandibular permanent posterior teeth with clinical signs indicative of irreversible pulpitis in patients with type 2 diabetes mellitus

Objectives-

1. To evaluate the clinical and radiographic success of complete pulpotomy in type 2 diabetic patients in permanent mandibular posterior teeth with clinical signs indicative of irreversible pulpitis.
2. To evaluate the clinical and radiographic success of root canal treatment in type 2 diabetic patients mandibular permanent posterior teeth with clinical signs indicative of irreversible pulpitis.

Population - Permanent mandibular posterior teeth with diagnosis of symptomatic irreversible pulpitis in patients with Type 2 Diabetes Mellitus.

Intervention/Treatment- complete pulpotomy

Comparator- Root canal treatment

Outcome- success of complete pulpotomy versus root canal treatment based on clinical and radiographic findings at 3, 6 and 12 months secondary outcome: assessment of quality of life 1 week, 6 and 12 months post treatment.

Time frame - 1 year

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus defined by HbA1c levels 6.5% - 8% OR FPG ≥126 mg/dL OR 2-hour plasma glucose ≥200 mg/dL during an OGTT OR A random plasma glucose of 200 mg/dL or higher in a patient with classic symptoms of hyperglycemia or hyperglycemic crisis
* Age between 18 - 70 years.
* Permanent mandibular posterior teeth with clinical and radiographic signs and symptoms indicative of irreversible pulpitis (PAI score ≤2)
* Tooth showing positive response to pulp sensibility testing with no tenderness on percussion.
* BMI<30 Kg/m2

Exclusion Criteria:

* Patients with immunocompromised diseases or chronic kidney disease
* Smokers, pregnant and lactating women
* Teeth with immature roots or retained deciduous tooth.
* Bleeding could not be controlled in ≥5 minutes.
* Tooth with signs and symptoms of apical periodontitis.
* Teeth with procedural errors, cracks, fractured teeth
* Tooth with probing depth more than 4mm.
* Positive history of antibiotic use in the past 1 month or requiring antibiotic prophylaxis and/or analgesic usage in past 3 days.
* Patients taking drugs that affect bone metabolism such as immune- suppressants, SSRIs, bisphosphonates, hormone replacement therapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
clinical success | 12 months
  Clinical success criteria No history of spontaneous pain or discomfort except for the initial days after treatment. No tenderness to palpation or percussion and the tooth is functional. Normal mobility and probing pocket depth. Soft tissues around tooth are normal with no swelling or sinus tract.
radiographic success | 12 months
  Radiographic success criteria No pathosis evident on the radiograph such as root resorption, furcal pathosis or new periapical pathosis. Periapical Index score 1 or 2

SECONDARY OUTCOMES:
quality of life assessment | 12 months
  OHRQoL assessment: OHIP-14 questionnare will be used to assess the quality of life. OHIP- 14 developed by Slade is a well-validated and reliable tool to assess OHRQoL. It consists of questionnaire in seven dimensions: functional limitation, physical pain, psychological discomfort, physical disability, psychological disability, social disability, and handicap. It will be scored using a Lickert scale: never=0; hardly ever=1; occasionally=2; fairly often=3; very often=4. Total score will be calculated ranging from 0-56, with higher score denoting the worst At the follow-up visits (1 week, 6 months, and 1 year), the patients will be reporting their responses after receiving the treatment by selecting from the following 3 options: the treatment will be improving the situation, the treatment will be worsening the situation, and no change will be being noticed

CONTACTS AND LOCATIONS:
Overall Officials: Jigyasa Duhan, MDS, Principal Investigator — PGIDS Rohtak
Locations (1):
- PGIDS Rohtak, Rohtak, Haryana, India